CLINICAL TRIAL: NCT00081510
Title: A Randomized Double-Blind Phase-2 Study of Anastrozole Plus Lonafarnib (SCH 66336) or Anastrozole Plus Placebo for the Treatment of Subjects With Advanced Breast Cancer
Brief Title: Anastrozole Plus Lonafarnib (SCH 66336) or Plus Placebo for the Treatment of Advanced Breast Cancer (P03480)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03480; NCT00098904 (obsolete NCT alias)
Record Dates: First submitted 2004-04-14; First posted 2004-04-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — lonafarnib; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lonafarnib plus Anastrozole (Experimental): Participants receive lonafarnib 200 mg orally (PO) twice per day (BID) beginning on Day 1 Cycle 1 and continuing until Progression of Disease, unacceptable toxicity, or other discontinuation criteria are met; and anastrozole 1 mg, PO, once per day (QD) for as long as the participant is receiving lonafarnib
  Interventions: Drug: Lonafarnib; Drug: anastrozole
- Placebo plus Anastrozole (Active Comparator): Participants receive placebo to lonafarnib PO BID beginning on Day 1 Cycle 1 until Progression of Disease, unacceptable toxicity, or other discontinuation criteria are met; and anastrozole, 1mg PO QD for as long as the participant is receiving placebo
  Interventions: Drug: Placebo; Drug: anastrozole

INTERVENTIONS:
Drug: Lonafarnib
  Other Names: SCH 66336
  Arms: Lonafarnib plus Anastrozole
Drug: Placebo
  Arms: Placebo plus Anastrozole
Drug: anastrozole

SUMMARY:
Primary Objective(s):

* To compare the activity (progression-free survival [PFS]) of anastrozole in combination with lonafarnib to that of anastrozole in combination with placebo in subjects with hormone-sensitive ADVANCED breast cancer.

Secondary Objective(s):

* To determine the effects of anastrozole in combination with lonafarnib on objective response, duration of response, overall survival, and safety in subjects with advanced breast cancer. To assess the exposure and pharmacokinetics of lonafarnib and anastrozole in the subject population.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who have histologically-confirmed breast cancer with the following characteristics:

  * estrogen and/or progesterone receptor positive,
  * locally advanced disease
  * distant metastatic disease, stage 4
* Subjects eligible for single-agent treatment with aromatase inhibitors for current disease.
* Subjects taking biophosphonates are allowed if they begin bisphosphonate therapy AT LEAST two weeks prior to randomization.
* Measurable disease (masses with clearly defined margins on radiological images and at least one diameter >=20 mm[>=10 mm if spiral CT]) or evaluable disease (masses with margins not clearly defined on radiological images or with no diameter >= 20 mm). Subjects with bone disease only are permitted if disease is evaluable.
* ECOG Performance Status of 0 or 1.
* Sufficient bone marrow reserve.
* Adequate hepatic and renal function: laboratory values within protocol requirements.

Exclusion Criteria:

* Subjects who have received more than one regimen of cytotoxic chemotherapy for advanced disease.
* Subjects with with CLINICALLY APPARENT brain metastases or extensive visceral disease, including extensive hepatic involvement or pulmonary lymphangitic spread of tumor.
* Subjects with prior treatments with FTIs.
* Subjects with a known or suspected hypersensitivity to any excipients in the lonafarnib formulation (Providone, Poloxamer 188, croscarmellose sodium, silicon dioxide, and magnesium stearate).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | When approximately 70 subjects have progressed

SECONDARY OUTCOMES:
Objective response rate (adjusted RECIST criteria), duration of response, and overall survival | When approximately 70 subjects have progressed
To access the exposure and pk of lonafarnib and anastrazole in the subject population. | When approximately 70 subjects have progressed